CLINICAL TRIAL: NCT04885036
Title: An RCT Study Investigating the Effectiveness of Emotion Focused Skills Training (EFST)
Brief Title: Effectiveness of Emotion Focused Skills Training (EFST)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Collaborators: South-Eastern Norway Regional Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SorlandetHF Zahl-Olsen
Record Dates: First submitted 2021-03-24; First posted 2021-05-13 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Mental Health Issue
Keywords: Emotion focused skills training; Treatment outcome; Effectiveness; Mental health
MeSH Terms: conditions — Psychological Well-Being | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: A Randomized Clinical Trial comparing Emotion-focused skills training (EFST) up against treatment as usual in an outpatient specialist mental health clinics family team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment As Usual (Active Comparator): This group will receive treatment as usual within the family unit
  Interventions: Behavioral: Treatment As Usual
- EFST intervention (Experimental): This group will receive an EFST stand alone treatment consisting of a two days EFST course and 6 individual parental guidance sessions
  Interventions: Behavioral: EFST intervention

INTERVENTIONS:
Behavioral: EFST intervention — EFST extended intervention is a stand-alone treatment that consist of a two days EFST group course followed by six weekly individual sessions of parental guidance by a licensed EFST therapist. The treatment is given indirectly to the child through work with the parent, thus it might remove or diminish the pressure on the children that suffer from mental health problems to solve their disorder themselves. In this condition a total of 19 hours of EFST treatment is provided.
  Arms: EFST intervention
Behavioral: Treatment As Usual — In the TAU condition, the families will receive treatment as usual that does not include EFST treatment. Recent research indicates that this is therapy of high quality carried out by highly qualified staff (Tilden et al., 2020; Zahl-Olsen et al., 2020).The therapists are educated psychologists, psychiatrist and family therapists. The TAU intends to be the best treatment for the child/ family based on the type of symptoms presented and requests from the patient and his/her family. We will measure the intensity and type of therapy given in this condition by information from the therapists and investigate that it did not include the main elements of EFST treatment.
  Arms: Treatment As Usual

SUMMARY:
Comparing the effectivity of an EFST parent supervision intervention against Treatment As Usual in an outpatient specialist health care clinics Family unit.

DETAILED DESCRIPTION:
The aim of this study is to compare two different treatment conditions and their effect on the mental health of children and adolescent clients.

The first condition is the typical mental health treatment offered when the family is motivated to receive family based interventions in the clinic, thus, treatment as usual TAU as provided by the cliniques family team. A prior study, including data from the same clinic, found that the TAU was associated with good outcomes, identifying effect sizes equal to what is usual in clinical studies

The second condition, labelled: EFST intervention is a parent guidance intervention delivered as a two-day intensive group course followed by six weekly guidance sessions for parents of children with mental health issues.

Both treatment conditions are currently delivered at the clinic and by randomly assigning clients to each of these we will be able to compare the effects they have on the mental health of children and adolescents. The results will possibly guide what treatments to offer in the future.

ELIGIBILITY:
Inclusion Criteria:

* Children with a wide range of diagnosis will be included.
* Children in the age group from 6-18 years in the mental health clinic will be invited to participate.
* It is preferred that both parents participate in the EFST treatment.

Exclusion Criteria:

* parents need to live with the child at least 50% of the time (if separated or divorced)
* Parents need to speak Norwegian to a degree that they can comprehend the psychoeducation and participate in the sessions without an interpreter.
* parents with ongoing substance abuse or mental states that make participation too difficult, e.g., psychosis, will be excluded.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2021-12-08 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-12-22 (Actual)

PRIMARY OUTCOMES:
Change in childrens symptoms and diagnosis | T0=At randomization, T1= 3 months after T0
  To establish and measure change in childrens symptoms and diagnosis of mental distress, our main outcome measure will be the semi-structured diagnostic interview Schedule for Affective Disorders and Schizophrenia, present and lifetime version (Kiddie-SADS-PL), DSM-IV version (Kaufman, 1997). the Kiddie-sads will be completed at randomization and then repeated after 3 months to investigate the presence of diagnosis. A diagnosis will be rated as present or not present, with the threshold for presence being defined as a score of at least 3 within each diagnosis.
Change in reported symptoms and distress | T0 = At randomization, T1 = 3 months after T0, T2 = 6 months after T0, T3 = 12 months after T0
  To measure change in childrens symptoms of mental distress, the Strength and Difficulties Questionnaire, SDQ (Goodman et al., 2000) will be used. The child will be filling it out him/herself electronically (from 11 yeas of age), as well as the parents and teacher. The SDQ consists of 25 items describing positive and negative attributes of children and adolescents that can be allocated to 5 subscales. Each item has to be scored on a 3-point scale with 0 = 'not true', 1 = 'somewhat true', and 2 = 'certainly true'. A total difficulties score will also be calculated(range 0-40).Lower scores indicates better outcome.

SECONDARY OUTCOMES:
Change in reported Health-Related Quality of Life | T0 = At randomization, T1 = 3 months after T0, T2 = 6 months after T0, T3 = 12 months after T0
  To measure change in self-perceived quality of life, the Health-Related Quality of Life KINDL-R is used (Bullinger et al., 2008). KINDL-R will be filled out by parent and child.The KINDL-R questionnaire comprises 24 items to which the respondents are asked to respond on a 5-point Likert scale (never, seldom, sometimes, often, all the time). The resulting subscales are physical well-being, emotional well-being, self-esteem, family, friends, and everyday functioning (school or nursery school/kindergarten). The subscales of these six dimensions can be combined to produce a total score. Sum scale scores will be calculated by summing up the answer scores (1-5) of each scale. All scales will be transformed so that values range from 0 to 100, with higher values representing better quality of life.
Changes in parents emotional style | T0 = At randomization, T1 = 3 months after T0, T2 = 6 months after T0, T3 = 12 months after T0
  To measure Changes in parents emotional style the Emotion-Related Parenting Styles, ERPS (Paterson et al., 2012) will be used. ERPS is self-report measure for parents. ERPS consists of 20 items. Each item has to be scored on a 5-point scale fram "always false" to "always true". Scores on the items draws four subscales: Emotion Coaching parenting style (EC), Parental Rejection of negative emotion (PR), Parental acceptance of negative emotion (PA), Feeling of uncertainty /ineffectiveness in emotion socialization (UI). Higher scores indicates a better outcome on sbscales: EC and PA. Lower scores indicates better outcome on subscales PR and UI.
Changes in parents emotion regulation | T0 = At randomization, T1 = 3 months after T0, T2 = 6 months after T0, T3 = 12 months after T0
  To measure Changes in parents emotion regulation the Difficulties in Emotion Regulation Scale, short-form, DERS-18 (Victor, S. E., & Klonsky, E. D. (2016) will be used. DERS is self-report measure for parents.The DERS-18 is comprised of three items per subscale, for six subscales (Awareness, Clarity, Goals, Impulse, Nonacceptance and Strategies), a total of 18 items. These include three reverse- coded items, all on the Awareness subscale. A total score can also be calculated. Lower scores indicates better outcome.
Change in parents symptoms mental distress | T0 = At randomization, T1 = 3 months after
  To measure mental health, and change in mental health in parents, the Hopkins Symptom Checklist-10 (HSCL-10) will be used. HSCL-10 is a self report form filled out by parents. It contains 10 items on a 4 point scale from 0=" Not at all" to 4="Very much". Higher scores indicates higher level of distress.HSCL-10 is a short form of the HSCL 25. A comparison study by Strand et al. showed that the shorter version of SCL performed almost as well as the full version. (Strand et al. 2003)
Change in the quality of parents relationship with child | T0 = At randomization, T1 = 3 months after T0, T2 = 6 months after T0, T3 = 12 months after T0
  To measure parents relationship with child, and changes in relationship with the child, "the relationship with child RWC" (Pinsof, 2017) will be used. RWC is a self report filled out by parents. It contains 6 items on a 5 point scale from "never" to "all the time". Higher scores indicates a better perceived relationship with the child.

CONTACTS AND LOCATIONS:
Overall Officials: Rune H Zahl-Olsen, Ph.D, Principal Investigator — Senior researcher at Sørlandet Hospital HF
Locations (1):
- Sørlandet Hospital HF, Kristiansand, Agder, Norway

IPD SHARING:
Plan to Share IPD: No
The data stems from a clinical population of vulnerable families

REFERENCES:
- [Derived] Severinsen L, Stiegler JR, Nissen-Lie HA, Shahar B, Zahl-Olsen R. Effectiveness of emotion focused skills training for parents: study protocol for a randomized controlled trial in specialist mental health care. BMC Psychiatry. 2022 Jul 7;22(1):453. doi: 10.1186/s12888-022-04084-x. PMID 35799120